CLINICAL TRIAL: NCT05219773
Title: A Comparison of Clinic-based Versus Home-based Spirometry.
Brief Title: Clinic Versus Home Spirometry
Acronym: COMPAIR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 288594
Record Dates: First submitted 2021-09-28; First posted 2022-02-02 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Asthma; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinic vs Home spirometry (Other): The collection of medical history and demographic data Spirometry testing in both the clinic and home setting. The measurement of height and weight. The evaluation of the perception of home spirometry via a survey.
  Interventions: Device: NuvoAir Air Next spirometer

INTERVENTIONS:
Device: NuvoAir Air Next spirometer — * The collection of medical history and demographic data
  * Spirometry testing in both the clinic and home setting.
  * The measurement of height and weight.
  * The evaluation of the perception of home spirometry via a survey.

SUMMARY:
The study aims to assess the differences between spirometry performed with the NuvoAir Air Next spirometer in the clinic setting with both direct and virtual supervision via a video call, and in the home setting with virtual supervision. This is will be achieved by comparing lung function values, specifically the FEV1 and FVC measurements. We also wish to evaluate participant's perceptions of home spirometry, by using a survey.

This is a multi-centre, cross-over study. The study will enrol participants with a diagnosis of asthma and COPD, across participating study sites until 68 have completed the study.

ELIGIBILITY:
Inclusion Criteria:

* An ability to provide fully informed consent.
* A diagnosis of asthma or COPD.
* Male or female aged ≥18 and ≤ 80 years of age.

Exclusion Criteria:

* Symptoms suggestive of COVID-19.
* An exacerbation of asthma or COPD or symptoms of a respiratory infection within the 30 days prior to the first visit.
* Any other clinically significant medical disease or uncontrolled concomitant disease, that is likely, in the opinion of the Investigator(s), to impact on the ability to participate in the study.
* The presence of any contraindications to spirometry.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2021-12-14 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
1. To compare spirometric values obtained from the NuvoAir Air Next device, directly supervised in clinic and virtually supervised in clinic and at home. | 8 days
  Over an 8-day period; the forced expiratory volume in 1 second (FEV1) and forced vital Capacity (FVC) will be measured at 4 points in the study over the 8 day study period. Twice in clinic and twice at home.
2. To compare spirometric values obtained from two virtually supervised tests performed at home, using the NuvoAir Air Next device. | 8 days
  The forced expiratory volume in 1 second (FEV1) and forced vital Capacity (FVC) will be measured via the NuvoAir Air Next spirometer at home at 2 points during the 8 day study period.

SECONDARY OUTCOMES:
To evaluate the participant's views of home spirometry via a survey. | 8 days
  A standardised survey to evaluate the participant's perception of home spirometry, will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Harrison, Principal Investigator — University of Nottingham
Locations (3):
- United Kingdom (3):
  - Respiratory Research Unit, Nottingham, Nottinghamshire
  - Bradford Teaching Hospitals NHS Foundation Trust, Bradford
  - The Rotherham NHS Foundation Trust, Rotherham

IPD SHARING:
Plan to Share IPD: No